CLINICAL TRIAL: NCT01990443
Title: A Randomized, Open-Label, Parallel-Group, Single-Dose Study to Characterize the Absolute Bioavailability of Reslizumab (220 mg) Following Subcutaneous Administration to Healthy Subjects
Brief Title: Absolute Bioavailability of Reslizumab in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: C38072/1107
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Absolute Bioavailability
Keywords: Reslizumab; monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reslizumab IV (Experimental): Reslizumab 220-mg administered Intravenously (IV)
  Interventions: Drug: Reslizumab IV
- Reslizumab SC (Experimental): Reslizumab 220-mg administered Subcutaneously (SC)
  Interventions: Drug: Reslizumab SC

INTERVENTIONS:
Drug: Reslizumab IV — Reslizumab 220-mg intravenous (IV)
  Arms: Reslizumab IV
Drug: Reslizumab SC — Reslizumab 220 mg administered subcutaneous (SC)
  Arms: Reslizumab SC

SUMMARY:
The primary objective of this study is to assess the absolute bioavailability of reslizumab following administration of a single subcutaneous (sc) dose to healthy non-Japanese participants

DETAILED DESCRIPTION:
The study is designed to assess the pharmacokinetics, safety and tolerability, immunogenicity, and pharmacodynamics of reslizumab

ELIGIBILITY:
Criteria for Inclusion: Subjects may be included in the study if they meet all of the following criteria:

All Subjects

1. Written informed consent is obtained.
2. The subject can read, speak, and write in English or Japanese (as applicable to the respective enrollment group).
3. The subject is in good health as determined by medical and psychiatric history, physical examination, brief neurologic examination, ECG, serum chemistry, hematology, urinalysis, and serology.
4. The subject, if a woman, is surgically sterile, 2 years postmenopausal, or, if of childbearing potential, is using a medically accepted method of contraception, and agrees to continued use of this method for the duration of the study and for 30 days after completion of the study. Acceptable methods of contraception include abstinence or an intrauterine device (known to have a failure rate of less than 1% per year).
5. The subject must be willing and able to comply with study restrictions and to remain at the clinic for the required duration at each visit. Non-Japanese Subjects
6. The subject has Caucasian parents and grandparents.
7. The subject is a man or woman 18 through 45 years of age with a body mass index (BMI) of 20.0 to 30.0 kg/m2, inclusive (Appendix A). Note: At least half of the subjects enrolled into each treatment group must be within the more stringent age and weight criteria noted below for Japanese subjects.

   Also, every effort should be made to enroll an approximately equal number of men and women.

   Japanese Subjects
8. The subject is a man or woman 20 through 45 years of age weighing 50 through 80 kg with a BMI of less than 28.0 kg/m2. Note: Every effort should be made to enroll an approximately equal number of men and women.
9. The subject was born in Japan.
10. The subject has Japanese parents and grandparents.
11. The subject has lived less than 5 years outside Japan.
12. The subject has a Japanese passport.
13. The subject has no plans to leave the US until at least 1 week after the end of the study.

Criteria for Exclusion: Subjects will be excluded from participating in this study if they meet 1 or more of the following criteria:

1. The subject has any clinically significant uncontrolled medical conditions (treated or untreated).
2. The subject has a clinically significant deviation from normal in ECG, physical examination, or brief neurologic examination findings, as determined by the investigator or the medical monitor.
3. The subject is a pregnant or lactating woman. (Any women becoming pregnant during the study will be withdrawn from the study.)
4. The subject has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery; a history of appendectomy is allowed).
5. The subject has received reslizumab in a previous study.
6. The subject has received an immunosuppressant drug or anti-interleukin-5 (anti-IL-5) antibody within 6 months before the dose of study drug.
7. The subject has received any investigational drug (non-biologic) within 30 days or 5 half-lives (whichever is longer) before the dose of study drug, or in the case of a new chemical entity, 3 months or 5 half-lives (whichever is longer) before the dose of study drug.
8. The subject has participated in any investigative biologics study within 6 months or 5 half-lives (whichever is longer) before the dose of study drug.
9. The subject has a known or suspected hypersensitivity or idiosyncratic reaction to anti-IL-5 antibodies, any compound present in the study drug, or monoclonal antibodies.
10. The subject has a history of any clinically important drug, vaccine and/or other allergies or there is indication of potential for allergic reactions. Pharmacokinetic Study-Healthy Subjects Clinical Study Protocol Study C38072/1107 8
11. The subject has received immunization with a live vaccine within 3 months prior to the dose of study drug or has immunization with a live or live attenuated vaccine planned within 3 months after the last dose of study drug.
12. The subject had or was suspected of having a parasitic infestation/infection within 6 months before the dose of study drug.
13. The subject has used any vitamins within 2 weeks before the dose of study drug or has used any systemic or topical prescription, or nonprescription (over-the-counter [OTC]) medication (except acetaminophen or ibuprofen) within 2 weeks or 5 half-lives (whichever is longer) before the dose of study drug.
14. The subject has used any herbal or nutritional supplements within 2 weeks before the dose of study drug.
15. The subject has donated blood or has a history of significant blood loss within 56 days prior to the dose of study drug.
16. The subject has donated plasma within 7 days prior to the dose of study drug.
17. The subject has, after resting for 5 minutes, elevated blood pressure (defined as seated systolic blood pressure of more than 140 mm Hg and/or seated diastolic blood pressure of more than 90 mm Hg), or low blood pressure (defined as seated systolic blood pressure of less than 90 mm Hg and/or seated diastolic blood pressure of less than 45 mm Hg). (Only 2 rechecks of the subject's blood pressure are permitted for eligibility purposes.)
18. The subject has, after resting for 5 minutes, a seated pulse of less than 45 or more than 90 beats per minute (bpm). (Only 2 rechecks of the subject's pulse are permitted for eligibility purposes.)
19. The subject has, within the past 2 years, habitually consumed more than 21 units of alcohol per week, or has a history of alcohol, narcotic, or any other substance abuse as defined by the Diagnostic and Statistical Manual of Mental Disorders of the American Psychiatric Association, Fourth Edition, Text Revision (DSM-IV-TR) (American Psychiatric Association 2000). Note: For the purpose of this study, a unit of alcohol is equal to 1 ounce of hard liquor, 5 ounces of wine, or 8 ounces of beer.
20. The subject has a positive urine drug screen (UDS) or alcohol test result.
21. The subject has a clinical laboratory test value(s) outside the range(s) specified below, or any other clinically significant laboratory abnormality as determined by the investigator or medical monitor:

    * hemoglobin value of less than 12 g/dL
    * aspartate aminotransferase (AST) or alanine aminotransferase (ALT) more than 2 times the upper limit of the normal range (ULN)
    * total bilirubin more than 25.7 μmol/L (1.5 mg/dL)
22. The subject has a positive test result for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or antibodies to hepatitis C.
23. The subject has, within 14 days before the dose of study drug, a clinically significant excessive consumption of coffee, tea, or other caffeine-containing beverages or food (ie, 600 mg/day of caffeine, 5 or more cups of coffee/day, or 10 or more cups of tea/day), or a combination of any of these beverages or foods.
24. The subject is a user or former user of nicotine-containing products (including but not limited to cigarettes, cigars, and chewing or dipping tobacco) who stopped use or consumption (ie, smoking, chewing, or pinching) of these nicotine-containing products less than 12 months before study drug administration or is using or has used topical or oral nicotine preparations for smoking cessation within the past 3 months before study drug administration.
25. The subject has had, within 4 weeks before the dose of study drug, a clinically significant illness, or within 1 week before the dose of study drug, any acute illness or, at screening or on the day before the first dose of study drug, has symptoms of any clinically significant or acute illness.
26. The subject has significant active infection (acute or chronic) within 4 weeks before the dose of study drug. aa. The investigator feels that the subject should not be enrolled in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Absolute bioavailability | From baseline to Day 140
  Absolute bioavailability calculated as (AUC0-∞)sc/(AUC0-∞)

SECONDARY OUTCOMES:
Maximum observed serum drug concentration (Cmax) | From baseline to Day 140
Time to maximum observed serum drug concentration (tmax) | From baseline to Day 140
AUC from time 0 to the time of the last measurable drug concentration (AUC0-t) | From baseline to Day 140
Percentage extrapolation | From baseline to Day 140
  Percentage extrapolation will be calculated as (AUC0-∞-AUC0-t)/(AUC0-∞)x100
Apparent serum terminal elimination rate constant (λz) | From baseline to Day 140
Associated elimination half-life (t½) | From baseline to Day 140
Total serum clearance (CL) | From baseline to Day 140
Volume of distribution (Vz) | From baseline to Day 140
Blood Eosinophils Levels | From baseline to Day 140
Anti-reslizumab antibodies | From baseline to Day 140
Summary of Participants with Adverse Events | From signing of consent form to Day 140
Blood samples for measurement of Anti-reslizumab antibodies | Baseline, days 14, 28, 84, 140
Area under the serum drug concentration by time curve from time 0 to infinity (AUC0-∞) | From baseline to Day 140

CONTACTS AND LOCATIONS:
Locations (1):
- Teva Investigational Site 10567, Anaheim, California, United States